CLINICAL TRIAL: NCT04233996
Title: Efficacy of Extended Infusion of β-lactam Antibiotics for the Treatment of Febrile Neutropenia in Haematologic Patients: a Randomised, Multicentre, Open-label, Superiority Clinical Trial (BEATLE)
Brief Title: Efficacy of Extended Infusion of β-lactam Antibiotics for the Treatment of Febrile Neutropenia in Hematologic Patients
Acronym: BEATLE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitari de Bellvitge (Other)
Collaborators: Institut d'Investigació Biomèdica de Bellvitge (Other); Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Carlota Gudiol, Principal Investigator, Hospital Universitari de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-001476-37
Record Dates: First submitted 2019-09-04; First posted 2020-01-21 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Febrile Neutropenia
Keywords: Febrile neutropenia; Beta-lactam antibiotics; Cefepime; Meropenem; Piperacillin-tazobactam; Extended infusion
MeSH Terms: conditions — Febrile Neutropenia | interventions — Piperacillin, Tazobactam Drug Combination; Cefepime; Meropenem

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Extended infusion (Experimental): Piperacillin-tazobactam, cefepime or meropenem will be administered in half time of the dosing interval
  Interventions: Drug: Piperacillin-Tazobactam 4 g-0.5 g; Drug: Cefepime 2000 mg; Drug: Meropenem 1000 mg
- Intermittent infusion (Active Comparator): Piperacillin-tazobactam, cefepime or meropenem will be administered in 30 minutes
  Interventions: Drug: Piperacillin-Tazobactam 4 g-0.5 g; Drug: Cefepime 2000 mg; Drug: Meropenem 1000 mg

INTERVENTIONS:
Drug: Piperacillin-Tazobactam 4 g-0.5 g — Patients with FN who empirical treatment with piperacillin-tazobactam 4g/6h
Drug: Cefepime 2000 mg — Patients with FN who required empirical treatment with cefepime 2g/8h
Drug: Meropenem 1000 mg — Patients with FN who required empirical treatment with meropenem 1g/8h

SUMMARY:
This study evaluates the administration of beta-lactam antibiotics in extended infusion in hematological patients with febrile neutropenia after 5 days of treatment. The beta-lactam antibiotics analyzed are the following: piperacillin-tazobactam, cefepime and meropenem. Half of patients will receive the antibiotic in intermittent infusion, while the other half will receive it in extended infusion.

DETAILED DESCRIPTION:
Febrile neutropenia (FN) is a very frequent complication in patients with hematological malignancies. It is associated with an important morbidity and mortality. Nowadays the use of betalactam antibiotics (BLA) in extended or continuous infusion (EI, CI) instead of intermittent infusion (II), has demonstrated a therapeutic success and lower mortality rate in critically ill intensive care patients. Neutropenic patients are a particular population since FN is assoicated with pathophysiological variations that compromise pharmacokinetic parameters of BLA, and may therefore, diminish their clinical efficacy. Information regarding the usefulness of BLA in EI in neutropenic hematologic patients is scarce.

The objective of this randomized clinical trial is to demonstrate the clinical superiority of the administration of BLA in EI compared to II in patients with FN.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (age ≥18 years) of both sexes.
2. Patients admitted in Hematological wards.
3. With any of the following diagnoses:

   1. Acute leukemia receiving chemotherapy.
   2. Autologous or allogeneic hematopoietic stem cell transplant recipients.
4. With an episode of febrile neutropenia: ≥ 38.0ºC and <500 neutrophils/mm3 or <1000 with a predicted decrease within 24-48 hours.
5. Patient requiring treatment with a beta-lactam antibiotic: cefepime, piperacillin /tazobactam or meropenem, in monotherapy or in combination with another antibiotic.
6. Written informed consent has been obtained from the patient or their legal representative grants.

Exclusion Criteria:

1. Allergy to study drugs.
2. Patient receiving systemic antibiotic treatment (except for prophylaxis) at the time of onset of febrile neutropenia.
3. Absence of fever.
4. Patients with epilepsy.
5. Severe renal impairment (defined as creatinine clearance <30 mL / min)
6. Previously enrolled patients in whom the time between the inclusion and the current episode is less than 5 weeks.
7. Previously enrolled patients without current resolution of the first episode.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-06-05 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical efficacy of extended infusion: Number of patients with defervescence | 5 days
  Number of patients with defervescence (<37.5 ºC, for 24 hours) without modifying the antibiotic treatment

SECONDARY OUTCOMES:
Pharmacokinetic target | 5 days
  Number of patients in whom the free antibiotic concentration remains above the MIC of the suspected or isolated microorganism, for 50%, 75% and 100% of the dosing interval.
Inflammatory biomarker | 5 days
  Number of patients who normalize or decrease in more than 50% of the peak value of the C-reactive protein.
Overall mortality at 30 days | 30 days
  Number of patients who died for any reason
Bacteraemia clearance | 30 days
  Time in days until bacteraemia clearance.
Adverse events | 30 days
  Incidence of adverse events in both groups
Pharmacokinetic analysis and population pharmacokinetics of meropenem, piperacillin and cefepime in neutropenic patients: Volume of distribution | 5 days
  Population mean value of volume of distribution of antibiotics during critical illness. Mean population volume of distribution will be derived from pooled data of antibiotic concentrations. Covariates of influence on volume of distribution will be incorporated within a population pharmacokinetic model.
Pharmacokinetic analysis and population pharmacokinetics of meropenem, piperacillin and cefepime in neutropenic patients: Clearance | 5 days
  Population mean value of clearance of antibiotics during critical illness. Mean population clearance will be derived from pooled data of antibiotic concentrations. Covariates of influence on drug clearance will be incorporated within a population pharmacokinetic model
Covariables analysis: biometric values: weight | 5 days
  Assessment of the impact of patient's weight [in kg]
Covariables analysis: biometric values: age | 5 days
  Assessment of the impact of patient's age [in years]
Covariables analysis: biochemical data: serum albumin | 5 days
  Assessment of the impact of total serum albumin [in g/L]
Covariables analysis: biochemical data: blood urea | 5 days
  Assessment of the impact of the urea [in mmol/L]
Covariables analysis: biochemical data: blood creatinine | 5 days
  Assessment of the impact of the creatinine [in umol/L]
Covariables analysis: clinical data: 24h diuresis | 5 days
  Assessment of the impact of 24h diuresis [in mL/day]
Pharmacokinetic analysis and population pharmacokinetics: time above a critical concentration value for plasma concentrations | 5 days
  Analysis of the antibiotic pharmacokinetic profiles by means of appropriate software to calculate the actual mean and median values of the fraction of the time between two successive drug administrations during which plasma concentrations of meropenem, piperacillin and cefepime remain above a critical value ("S" breakpoint of the corresponding antibiotic [meropenem, piperacillin and cefepime: European Committee for Antimicrobials Susceptibility Testing [EUCAST] value) in the study population, and to determine its value in a simulated population (Monte Carlo simulations; 1000 simulated patients).

CONTACTS AND LOCATIONS:
Overall Officials: Carlota Gudiol, PhD, Principal Investigator — Hospital Universitari de Bellvitge
Locations (1):
- Hospital Duran i Reynals, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Laporte-Amargos J, Gudiol C, Arnan M, Puerta-Alcalde P, Carmona-Torre F, Huguet M, Albasanz-Puig A, Parody R, Garcia-Vidal C, Del Pozo JL, Batlle M, Tebe C, Rigo-Bonnin R, Munoz C, Padulles A, Tubau F, Videla S, Sureda A, Carratala J. Efficacy of extended infusion of beta-lactam antibiotics for the treatment of febrile neutropenia in haematologic patients: protocol for a randomised, multicentre, open-label, superiority clinical trial (BEATLE). Trials. 2020 May 18;21(1):412. doi: 10.1186/s13063-020-04323-0. PMID 32423462
- See also: Spanish clinical trial registration (REEC, registro español de estudios clínicos) — https://reec.aemps.es/reec/public/detail.html